CLINICAL TRIAL: NCT01344421
Title: Movement Pattern in Patients With Hip Dysplasia Operated With Minimally Invasive Approach in Peri-acetabular Osteotomy (PAO)
Brief Title: Movement Pattern in Patients With Hip Dysplasia
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Other Study IDs: M-20100206
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Hip Dysplasia
Keywords: Movement capture system; Movement analysis; Hip dysplasia; Hip pain; Quality of life; Physical function
MeSH Terms: conditions — Hip Dislocation | interventions — Polyamine Oxidase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- hip dysplasia: Patients with hip dysplasia
  Interventions: Procedure: Minimally invasive approach for Periacetabular osteotomy
- Healthy people: Enrolled from the patients acquaintance circle

INTERVENTIONS:
Procedure: Minimally invasive approach for Periacetabular osteotomy — A peri-acetabular osteotomy is a surgery performed to correct the dysplastic acetabulum and reduce joint contact pressures and early osteoarthritis.
  Other Names: PAO (periacetabular osteotomy)
  Groups: hip dysplasia

SUMMARY:
The purpose of this study is to examine the movement pattern in patients with hip dysplasia preoperative, six and 12 month after minimally invasive approach for Periacetabular osteotomy (PAO). Secondary to examine the movement pattern in patients compared to healthy controls and historical data.

DETAILED DESCRIPTION:
Congenital hip dysplasia is a disease characterised by pathological changes in the hip joint. Hip dysplasia is a normal disease with a prevalence of 4.3% in men and 3.6 in woman. Untreated hip dysplasia is a known cause of developing osteoarthritis early in life and symptoms as pain, hip instability together with a changed gait pattern are normal. Symptomatic hip dysplasia is seen in patients between 15 and 55 years and can be unilateral as well as bilateral. Causes of hip dysplasia are described as genetic, mechanic or hormonal.

Today patients with hip dysplasia are offered a hip conserving surgery before the osteoarthritis has developed. In 2003 a minimally invasive approach for periacetabular osteotomy (PAO) was introduced at Aarhus University Hospital. An advantage of minimally invasive approach compared to the classical Bernese periacetabular osteotomy is minimal impact of the soft tissues in the hip region.

Hip pain and activity limitations highly affect quality of life and physical function. The gait distance is reduced and patients have to compensate to relieve the pressure on the hip joint. Knowledge about the dynamics of the gait and running pattern in patients with dysplasia is important to understand the consequences of the dysplastic hip joint. Furthermore knowledge about gait compensations is relevant for the clinicians in the management and treatment of patients with hip dysplasia.

Today, gait and running compensation is unknown after minimally invasive approach The purpose of this study is, therefore, to examine the movement pattern in patients with hip dysplasia preoperative, six and 12 month after minimally invasive approach for Peri-acetabular osteotomy (PAO). Secondary to examine the movement pattern in patients compared to healthy controls and historical data.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hip dysplasia
* Patients in the age of 18-60 years
* Patients, who can speak, understand and read Danish

Exclusion Criteria:

* Persons with hip dysplasia secondary to other hip conditions such as Calvé Perthes and epiphysiolysis.
* Persons who have had alloplastic surgery in the hip, knee or ankle.
* Persons with diseases that affect the gait pattern.
* Persons with serious hip, knee, ankle or back pain.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients diagnosed with hip dysplasia and waiting for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Hip flexion's muscle moment in stance evaluated in gait, run and jump test | Preoperative (baseline), 6 and 12 month postoperative
  Examined using 3D Movement Capture System

SECONDARY OUTCOMES:
Hip extension angle evaluated in gait, run and jump test | Preoperative (baseline), 6 and 12 month postoperative
  Examined using 3D Movement Capture Systen
On-set of the hip muscles evaluated in gait, run and jump test | Preoperative (baseline), 6 and 12 month postoperative
  Examined using skin electromyography (EMG)
Function, sports and recreational activities | Preoperative (baseline), 6 and 12 month postoperative
  Evaluated with Hip Dysfunction and Osteoarthritis Outcome Score (HOOS) and The Copenhagen Hip and Groin Outcome Score (HAGOS)
Quality of life | preoperative (baseline), 6 and 12 month postoperative
  Evaluated with Hip Dysfunction and Osteoarthritis Outcome Score (HOOS) and The Copenhagen Hip and Groin Outcome Score (HAGOS)

CONTACTS AND LOCATIONS:
Overall Officials: Julie S Jacobsen, MSc, Principal Investigator — Aarhus University Hospital; Inger Mechlenburg, MSc, PhD, Principal Investigator — Aarhus University Hospital; Kjeld Søballe, Prof. Dr.med, Study Chair — Aarhus University Hospital; Henrik Sørensen, PhD, Study Chair — University of Aarhus; Dennis Nielsen, MSc, Study Chair — University of Aarhus
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Sorensen H, Skalshoi O, Nielsen DB, Jacobsen JS, Soballe K, Mechlenburg I. Hip muscle and joint contact forces before, 6 and 12 months after minimally invasive periacetabular osteotomy. Hip Int. 2021 Sep;31(5):676-682. doi: 10.1177/1120700020925411. Epub 2020 May 4. PMID 32366122